CLINICAL TRIAL: NCT06457555
Title: Intensive Care Nurses' Knowledge Levels and Experiences Regarding Pressure Sore Prevention: Mixed Method
Brief Title: Knowledge Levels and Experiences of Intensive Care Nurses on the Prevention of Pressure Sores: Mixed Method
Status: Active, not recruiting | Type: Observational
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Doctor Lecturer Ayşe UÇAK, assistant professor AYŞE UÇAK, Burdur Mehmet Akif Ersoy University
Other Study IDs: AYŞEUÇAK; GO 2023/568 (Other: Ethics Committee)
Record Dates: First submitted 2024-03-30; First posted 2024-06-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Nurses; Pressure Ulcer; Critical Care
Keywords: Intensive Care Nurse; pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nurses working in adult intensive care units: In the research, parallel data type was used in the convergent parallel mixed design (convergent parallel) in order to obtain meticulous, valid and reliable data through survey questions and individual interviews. In the quantitative dimension of the research, nurses working in internal medicine, neurology, cardiology and surgical intensive care clinics of a public hospital were examined.
  While determining their level of knowledge regarding the prevention of pressure ulcers, it is also aimed to determine their experiences regarding practices to prevent pressure ulcers in a qualitative dimension.
  Interventions: Other: type of parallel data in a convergent parallel hash pattern (near time)

INTERVENTIONS:
Other: type of parallel data in a convergent parallel hash pattern (near time) — This study is a mixed method research conducted to determine the knowledge levels and experiences of nurses working in adult intensive care units regarding the prevention of pressure sores. In accordance with the purpose of the study, parallel data type in convergent parallel mixed design will be used as the research design. The quantitative phase will be conducted as a descriptive survey, and the qualitative phase will be conducted as a descriptive case study design. In this mixed design, equal priority, parallel timing and combining results during interpretation are planned.

SUMMARY:
This research aims to determine the knowledge levels and practices of intensive care nurses regarding the prevention of pressure sores.

The main questions it aims to answer are:

1. What is the level of knowledge of intensive care nurses regarding the prevention of pressure sores?
2. What is the impact of sociodemographic characteristics of intensive care nurses on their knowledge level regarding the prevention of pressure sores?
3. What are the experiences of intensive care nurses regarding their practices for the prevention of pressure sores? In this research, a survey and interview technique will be applied to determine the knowledge levels and experiences of nurses working in adult intensive care units regarding the prevention of pressure sores and their practices.

DETAILED DESCRIPTION:
This study is a mixed method research conducted to determine the knowledge levels and experiences of nurses working in adult intensive care units regarding the prevention of pressure sores. In accordance with the purpose of the study, parallel data type in convergent parallel mixed design will be used as the research design. The quantitative phase will be conducted as a descriptive survey, and the qualitative phase will be conducted as a descriptive case study design. In this mixed design, equal priority, parallel timing and combining results during interpretation are planned. The research will be conducted with nurses working in adult intensive care units of a public hospital located in a city center. 'Sociodemographic Form', 'Pressure Ulcer Knowledge Level Assessment Tool 2.0- Updated Version', 'Semi-Structured Interview Form' will be used as data collection tools. Within the scope of our research questions, quantitative and qualitative data will be analyzed independently of each other. In the discussion section, the integration of quantitative and qualitative evidence will be interpreted by making analytical generalization by combining data without transformation.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in adult intensive care units Agreeing to participate in the research

Exclusion Criteria:

* Nurses who do not work in adult intensive care units Nurses who did not agree to participate in the research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the research consists of nurses working in adult intensive care clinics of a public hospital. At the quantitative stage, an attempt will be made to reach the universe. In the qualitative phase of the research, intensive care nurses who agreed to be interviewed during the collection of quantitative data will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure Ulcer Knowledge Level of Intensive Care Nurses | four months
  Pressure Ulcer Knowledge Level Assessment Tool 2.0-Updated Version (PUKAT 2.0): The Turkish adaptation of the PUKAT 2.0 measurement tool was made by Dallı et al. (2021). PUKAT 2.0 is a measurement/test tool scored as multiple choice true-false. It consists of a total of 25 questions. It is scored according to the number of correct answers given by the individual. The Cronbach Alpha value of the internal consistency reliability of the measurement tool was found to be 0.72. All results will be coded as binary variables: correct (1) and incorrect (0). If the answer is not known, more than one answer or no answer is selected, the result will be coded as incorrect. The total score for each participant will be calculated as the sum of the correct answers. The minimum score to be obtained from the scale is 0 and the maximum score is 25. As the scores increase, the level of knowledge increases.
Intensive Care Nurses' experiences | four months
  The qualitative data obtained from the research will be evaluated with inductive content analysis. In order to increase the validity of the data, two researchers will examine the transcripts separately and comprehensive readings will be made. Codes will be created and compared by interpreting them in terms of differences and similarities, categories and sub-themes will be obtained. Main themes and sub-themes will be determined and research objectives will be tried to be given within the framework of the pattern between the interviews.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE UÇAK, Principal Investigator — Mehmet Akif Ersoy University
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided